CLINICAL TRIAL: NCT00900354
Title: Pharmacokinetics of Actinomycin D in Children With Cancer
Brief Title: Pharmacokinetics of Dactinomycin in Young Patients With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CCLG-PK-2006-07; CDR0000531136 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2005-002996-34; EU-20643; CCLG-CTA-21275/0218/001-0001
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Genetic Testing; Mass Spectrometry

INTERVENTIONS:
Genetic: molecular genetic technique
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer receiving dactinomycin may help doctors learn how dactinomycin works in the body and how patients will respond to treatment.

PURPOSE: This laboratory study is evaluating the pharmacokinetics of dactinomycin in young patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics (PKs) of dactinomycin in pediatric patients with cancer.
* Determine the degree of interpatient variation in the PKs of this drug.
* Determine the influence of characteristics such as age, tumor type, and concurrent therapy on drug PKs in these patients.
* Correlate drug PKs with clinical response and toxicity observed in these patients, focusing particularly on the incidence of severe liver toxicity or veno-occlusive disease.
* Correlate pharmacogenetic variability with clinical and PK data.

OUTLINE: This is a multicenter study.

Patients undergo blood collection for pharmacokinetic sampling of dactinomycin at baseline (prior to the initiation of dactinomycin) and periodically during course 1 of chemotherapy. An additional blood sample is obtained before or after treatment for the collection of peripheral blood lymphocytes. DNA from these cells is isolated and investigated for genetic variation in genes relevant to the pharmacology of dactinomycin. Plasma concentrations of dactinomycin are determined by liquid chromatography mass spectrometry analysis.

Patients are followed for 2 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Currently being treated with dactinomycin on a clinical trial at a United Kingdom Children's Cancer Study Group center

PATIENT CHARACTERISTICS:

* Single- or double-lumen central venous catheter or portacath in place

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Pharmacokinetics (PKs) of dactinomycin
Degree of interpatient variation of drug PKs
Influence of characteristics such as age, tumor type, and concurrent therapy on drug PKs
Correlation of drug PKs with clinical response and toxicity, particularly the incidence of severe liver toxicity or veno-occlusive disease

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Veal, Study Chair — University of Newcastle Upon-Tyne; Alan Boddy, PhD — University of Newcastle Upon-Tyne
Locations (22):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - University of Newcastle-Upon-Tyne Northern Institute for Cancer Research, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Kim HY, Veal GJ, Zhou F, Boddy AV. The role of solute carrier (SLC) transporters in actinomycin D pharmacokinetics in paediatric cancer patients. Eur J Clin Pharmacol. 2018 Dec;74(12):1575-1584. doi: 10.1007/s00228-018-2544-z. Epub 2018 Aug 30. PMID 30167756